CLINICAL TRIAL: NCT02093390
Title: A Phase 1, Open-Label, Drug-Drug Interaction Study to Evaluate the Effects of Multiple Oral Doses of Fluconazole and Atorvastatin on the Pharmacokinetics of a Single Oral Dose of TAK-385 in Healthy Subjects
Brief Title: A Phase 1 Study to Evaluate the Effects of Fluconazole and Atorvastatin on the Pharmacokinetics of TAK-385 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C27005; U1111-1183-0138 (Registry Identifier: WHO)
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer; Endometriosis
MeSH Terms: conditions — Prostatic Neoplasms; Endometriosis | interventions — relugolix; Fluconazole; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-385 + fluconazole (Experimental): TAK-385 40 mg, tablet, orally once on Day 1 and fluconazole 400 mg, tablet, orally on Day 6 then 200 mg, tablet, orally once daily on Days 7 to 9 followed by a single dose of TAK-385 in combination with fluconazole 200 mg on Day 10 then fluconazole 200 mg, tablet, orally once daily alone on Days 11 to 14.
  Interventions: Drug: TAK-385; Drug: Fluconazole
- TAK-385 + atorvastatin (Experimental): TAK-385 40 mg, tablet, orally once on Day 1 and atorvastatin 80 mg, tablet, orally once daily on Days 6 to 9 followed by a single dose of TAK-385 in combination with atorvastatin 80 mg on Day 10 then atorvastatin 80 mg, tablet, orally once daily alone on Days 11 to 14.
  Interventions: Drug: TAK-385; Drug: Atorvastatin

INTERVENTIONS:
Drug: TAK-385 — TAK-385 tablets
Drug: Fluconazole — Fluconazole tablets
  Arms: TAK-385 + fluconazole
Drug: Atorvastatin — Atorvastatin tablets
  Arms: TAK-385 + atorvastatin

SUMMARY:
This is a nonrandomized, open-label, fixed-sequence, 2-arm study designed to assess the effect of multiple doses of fluconazole or atorvastatin on the single-dose pharmacokinetics of TAK-385 in healthy adult subjects.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-385. TAK-385 was being tested to assess if the way it is processed the body changes when it administered with other medications (fluconazole or atorvastatin). This study looked at lab results in people who took TAK-385.

The study enrolled 40 patients. Participants were assigned to one of the two treatment groups:

* TAK-385 40 mg and fluconazole 400 mg on Day 6 and 200 mg on Days 7 to 14
* TAK-385 40 mg and atorvastatin 80 mg on Days 6-14

Participants in the fluconazole arm were administered TAK-385 on Days 1 and 10 and fluconazole on Days 6 through 14. Participants in the atorvastatin arm were administered TAK-385 on Days 1 and 10 and atorvastatin on Days 6 through 14.

This single-center trial was conducted in the United States. The overall time to participate in this study was 4 weeks. Participants made multiple visits to the clinic, including one 16-day period of confinement to the clinic, and a final visit 7 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria

Each subject must meet all the following inclusion criteria to be enrolled in the study:

1. Age 18 to 55 years, inclusive, at the time of consent.
2. Healthy adult male or female in good health, as determined by a physician evaluation
3. Weight ≥ 45 kg and body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive, at screening.
4. Nonsmoker and does not use tobacco-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, or nicotine patch or gum).

Exclusion Criteria Subjects meeting any of the following exclusion criteria are not to be enrolled in the study.

1. The subject has a history of drug abuse (defined as any illicit drug use) within 1 year before screening or is unwilling to abstain from drugs throughout the study.
2. The subject is unwilling to agree to abstain from caffeine and alcohol-containing products from 72 hours before check-in (Day -1) to completion of the final assessment.
3. The subject has taken any prescription medicine or herbal preparations (eg, St John's wort) or received any immunizations within 30 days before check-in (Day -1).
4. The subject has taken any over the counter (OTC) medications or vitamin supplements within 14 days before check-in (Day -1). The subject is unwilling to agree to abstain from consumption of grapefruit or grapefruit-containing products from 72 hours before check-in (Day -1) to completion of the final assessment.
5. The subject has current or recent (within 6 months) history of gastrointestinal disease that would be expected to influence the absorption of drugs.
6. The subject has a positive test result for hepatitis B surface antigen, hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody or antigen, or serological reactions for syphilis at screening.
7. The subject has a clinically significant ECG abnormality at screening or check-in (Day -1) or a QTc interval (by Fridericia's correction) of 450 msec or greater, or the subject has a history of cardiac disease.
8. The subject has abnormal laboratory values suggesting a clinically significant disease at screening or check-in (Day -1) .
9. Female subjects who are lactating and breastfeeding or pregnant before the first dose of study drug.
10. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in the United States from 13 March 2014 to 19 April 2014
Pre-assignment Details: Healthy participants were enrolled equally in 1 of 2 treatment groups: TAK-385 + fluconazole or TAK-385 + atorvastatin.
Period: Overall Study
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- TAK-385 + Fluconazole: TAK-385 40 mg, tablet, orally once on Day 1 and fluconazole 400 mg, tablet, orally on Day 6 then 200 mg, tablet, orally once daily on Days 7 to 9 followed by a single dose of TAK-385 in combination with fluconazole 200 mg on 10 day then fluconazole 200 mg, tablet, orally once daily alone on Days 11 to 14.
- TAK-385 + Atorvastatin: TAK-385 40 mg, tablet, orally once on Day 1 and atorvastatin 80 mg, tablet, orally once daily on days 6 to 9 followed by a single dose of TAK-385 in combination with atorvastatin 80 mg on 10 day then atorvastatin 80 mg, tablet, orally once daily alone on Days 11 to 14.
- Total: Total of all reporting groups
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (9.74) | 40.2 (9.71) | 38.8 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Black or African American | 2 | 3 | 5
  White | 18 | 16 | 34
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 16 | 15 | 31
  Not Hispanic or Latino | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Weight [Mean (Standard Deviation); unit: kg] | 70.77 (9.137) | 71.96 (12.693) | 71.36 (10.933)
Height [Mean (Standard Deviation); unit: cm] | 163.6 (11.51) | 163.3 (12.10) | 163.4 (11.65)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.466 (2.296) | 26.567 (2.838) | 26.516 (2.548)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration of TAK-385 on Day 1
Description: Cmax is the peak concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 1 (Predose and multiple time points up to 120 hours postdose)
Population: Pharmacokinetic (PK)-Evaluable population included all enrolled participants who received at least one dose of study drug and had data available for analysis of the PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 20 | 20
ng/mL | 10.9 (9.34) | 20.1 (15.1)

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration of TAK-385 on Day 10
Description: as for outcome 1
Time Frame: Day 10 (Predose and multiple time points up to 120 hours postdose)
Population: PK-Evaluable population included all enrolled participants who received at least one dose of study drug and had data available for analysis of the PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 19 | 19
ng/mL | 14.4 (10.7) | 14.1 (8.41)

3. Primary Outcome: AUC(0-tlast): Area Under the Plasma Concentration Curve From Time Zero to the Time of the Last Quantifiable Concentration of TAK-385 on Day 1
Description: Area under the plasma concentration versus time curve from zero to the time of the last quantifiable concentration.
Time Frame: Day 1 (Predose and multiple time points up to 120 hours postdose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 20 | 19
ng*hr/mL | 87.4 (38.1) | 116.0 (56.3)

4. Primary Outcome: AUC(0-tlast): Area Under the Plasma Concentration Curve From Time Zero to the Time of the Last Quantifiable Concentration of TAK-385 on Day 10
Description: Area under the plasma concentration versus time curve from zero to the time of the last quantifiable concentration.
Time Frame: Day 10 (Predose and multiple time points up to 120 hours postdose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 19 | 19
ng*hr/mL | 104.0 (40.5) | 99.8 (31.2)

5. Primary Outcome: AUC(0-inf): Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity of TAK-385 on Day 1
Description: Area under the plasma concentration-time curve from time 0 to infinity.
Time Frame: Day 1 (Predose and multiple time points up to 120 hours postdose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 20 | 19
ng*hr/mL | 92.6 (40.2) | 123.0 (59.6)

6. Primary Outcome: AUC(0-inf): Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity of TAK-385 on Day 10
Description: Area under the plasma concentration-time curve from time 0 to infinity.
Time Frame: Day 10 (Predose and multiple time points up to 120 hours postdose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 19 | 19
ng*hr/mL | 112.0 (43.4) | 108.0 (32.3)

7. Secondary Outcome: Number of Participants With at Least 1 Treatment Emergent Adverse Event (AE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: First dose of study drug through the end of the study (22 days ± 3 days)
Population: Safety population included all randomized participants with at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 20 | 20
participants | 5 | 6

8. Secondary Outcome: Number of Participants With Clinical Significant Changes in Vital Signs
Description: Vital sign measurements included oral temperature, heart rate, supine (after 3 to 5 minutes in this position) and standing (after 3 to 5 minutes in this position) measurements of diastolic and systolic blood pressure.
Time Frame: Baseline and First dose of study drug through the end of the study (22 days ± 3 days)
Population: Safety population included all randomized participants with at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 20 | 20
participants | 0 | 0

9. Secondary Outcome: Number of Participants With Clinical Significant Changes in Electrocardiogram (ECG) Findings
Description: A 12-lead ECG was administered on Days 1,9,10,11,15.
Time Frame: Baseline and First dose of study drug through Day 15
Measure: Number; unit: participants
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 20 | 20
participants | 0 | 0

10. Secondary Outcome: Number of Participants With Clinical Significant Changes in Laboratory Tests
Description: Blood samples were collected for analysis of clinical chemistry and hematological parameters and urine samples were obtained for urinalysis. Clinical laboratory evaluations were performed at central and /local laboratories.
Time Frame: Baseline and First dose of study drug through the end of the study (22 days ± 3 days)
Population: Safety population included all randomized participants with at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 20 | 20
participants | 0 | 0

11. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration of TAK-385
Description: Tmax is the time to reach the maximum concentrations (Cmax), equal to time (hours) to Cmax.
Time Frame: Days 1 and 10 (Predose and multiple time points up to 120 hours postdose)
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 20 | 20
hours
  Day 1 (n=20, 20) | 1.00 [0.50 to 6.00] | 1.00 [0.492 to 2.01]
  Day 10 (n=19, 19) | 1.00 [0.499 to 6.01] | 1.01 [0.501 to 4.02]

12. Secondary Outcome: AUC (0-120): Area Under the Plasma Concentration-Time Curve From Time 0 to 120 Hours of TAK-385
Description: Area under the plasma concentration versus time curve from 0 to 120 hours after study drug administration.
Time Frame: Days 1 and 10 (Predose and multiple time points up to 120 hours postdose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 20 | 19
ng*hr/mL
  Day 1 (n=20,19) | 87.4 (38.1) | 116.0 (56.3)
  Day 10 (n=19,19) | 104.0 (40.5) | 99.8 (31.2)

13. Secondary Outcome: Terminal Disposition Half-life (t1/2) of TAK-385
Description: Terminal disposition half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: Days 1 and 10 (Predose and multiple time points up to 120 hours postdose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 20 | 19
hours
  Day 1 (n=20, 19) | 34.8 (3.38) | 36.5 (3.74)
  Day 10 (n=19, 19) | 39.2 (3.57) | 41.1 (5.11)

14. Secondary Outcome: Apparent Total Body Clearance (CL/F) of TAK-385
Time Frame: Days 1 and 10 (Predose and multiple time points up to 120 hours postdose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 20 | 19
liters/hour
  Day 1 (n=20, 19) | 502 (189) | 420 (244)
  Day 10 (n=19, 19) | 421 (186) | 406 (144)

15. Secondary Outcome: Fraction Excreted Unchanged (Fe) of TAK-385
Description: Fraction of TAK-385 excreted in the urine unchanged.
Time Frame: Days 1 and 10 (Predose and multiple time points up to 120 hours postdose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent of TAK-385
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Number analyzed (Participants) | 20 | 19
percent of TAK-385
  Day 1 (n=20, 19) | 1.56 (0.720) | 1.99 (1.17)
  Day 10 (n=20, 19) | 1.61 (0.813) | 1.40 (0.426)

16. Secondary Outcome: Plasma Trough Concentrations for Fluconazole
Description: Blood samples for fluconazole trough levels were collected predose (before dosing with fluconazole and before breakfast) on Days 8 through 12.
Time Frame: Days 8 to 12 Predose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-385 + Fluconazole
Number analyzed (Participants) | 20
ng/mL
  Day 8 | 6330 (1100)
  Day 9 | 6540 (1180)
  Day 10 | 7030 (1270)
  Day 11 | 7030 (1540)
  Day 12 | 7200 (1560)

17. Secondary Outcome: Plasma Trough Concentrations for Atorvastatin
Description: Blood samples for atorvastatin trough levels were collected predose (before dosing with atorvastatin and before breakfast) on Days 8 through 12.
Time Frame: Days 8 to 12 Predose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-385 + Atorvastatin
Number analyzed (Participants) | 19
ng/mL
  Day 8 | 0.742 (0.444)
  Day 9 | 0.753 (0.351)
  Day 10 | 0.702 (0.385)
  Day 11 | 0.559 (0.263)
  Day 12 | 0.536 (0.203)

ADVERSE EVENTS:
Time Frame: Up to 25 days
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-385 + Fluconazole | TAK-385 + Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/20 | 6/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-385 + Fluconazole (N=20) | TAK-385 + Atorvastatin (N=20)
Application site dermatitis (General disorders) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.